CLINICAL TRIAL: NCT06555913
Title: Maitland Mobilization and Scapular Stabilization Exercises on Shoulder Dysfunction Post Neck Dissection Surgeries
Brief Title: Maitland Mobilization and Scapular Stabilization Shoulder Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Mamdouh Abd-Elsalam Shaaban, Specialist of Physical Therapy - Hosh Essa Hospital - El-Behira., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 81893
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer
Keywords: Maitland Mobilization; Scapular Stabilization; Shoulder Dysfunction; Neck Dissection Surgeries
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Maitland Mobilization and Scapular Stabilization (Experimental): This group included twenty patients suffering from shoulder disability following NDS (modified radical, selective). They received Maitland mobilization Technique and scapular stabilization exercises in addition to the traditional physical therapy program which included (ROM exercises, stretching exercises and strengthening exercises for shoulder muscles) 3 sessions per week, for 2 months.
  Interventions: Other: Maitland Mobilization; Other: Scapular Stabilization; Other: Traditional Physical Therapy
- Maitland Mobilization (Experimental): This group included twenty patients suffering from shoulder disability following NDS (modified radical, selective). They received Maitland mobilization Technique in addition to the traditional physical therapy program which included (ROM exercises, stretching exercises and strengthening exercises for shoulder muscles) 3 sessions per week, for 2 months.
  Interventions: Other: Maitland Mobilization; Other: Traditional Physical Therapy
- Scapular Stabilization (Experimental): This group included twenty patients suffering from shoulder disability following NDS (modified radical, selective). They received scapular stabilization exercises in addition to the traditional physical therapy program which include (ROM exercises, stretching exercises and strengthening exercises for shoulder muscles) 3 sessions per week, for 2 months.
  Interventions: Other: Scapular Stabilization; Other: Traditional Physical Therapy

INTERVENTIONS:
Other: Maitland Mobilization — MM applies a passive oscillatory technique, classified from Grade I-IV with respect to intensity, to the shoulder in order to treat pain and stiffness.
  Grade I refers to an intensity of small amplitude that is applied at the beginning of the joint ROM, where there is no loading on connective tissue; it is often used in cases of severe pain
  Arms: Maitland Mobilization; Maitland Mobilization and Scapular Stabilization
Other: Scapular Stabilization — Scapular stabilization exercises are thought to have an important role in improving pain and dysfunction in the shoulder. The concept that an unstable
  scapula is associated with pathology and dysfunction of the shoulder is well accepted. The predominant theory emphasizes that for optimal function of the glenohumeral joint, the scapula must provide a stable base upon which upper extremity tasks are completed. Impaired scapular stability increases the risk for pathologies such as impingement or rotator cuff tears
  Arms: Maitland Mobilization and Scapular Stabilization; Scapular Stabilization
Other: Traditional Physical Therapy — ROM exercises, stretching exercises and strengthening exercises for shoulder muscles

SUMMARY:
Sixty patients from both genders suffering from shoulder disability post unilateral NDS (modified radical, selective) will participate in this study. Their ages will be ranged from 30 to 50 years. They will be selected randomly from Damanhur Oncology center, El-Behira, Egypt. They will be randomly distributed into three equal groups (each group 20 patients).

DETAILED DESCRIPTION:
Design of the study:

In this study the patients were randomly assigned into three equal groups (twenty patients for each group).

Group (A) :

This group included twenty patients suffering from shoulder disability following NDS (modified radical, selective). They received Maitland mobilization Technique and scapular stabilization exercises in addition to the traditional physical therapy program which included (ROM exercises, stretching exercises and strengthening exercises for shoulder muscles) 3 sessions per week, for 2 months.

Group (B):

This group included twenty patients suffering from shoulder disability following NDS (modified radical, selective). They received Maitland mobilization Technique in addition to the traditional physical therapy program which included (ROM exercises, stretching exercises and strengthening exercises for shoulder muscles) 3 sessions per week, for 2 months.

Group (C) :

This group included twenty patients suffering from shoulder disability following NDS (modified radical, selective). They received scapular stabilization exercises in addition to the traditional physical therapy program which include (ROM exercises, stretching exercises and strengthening exercises for shoulder muscles) 3 sessions per week, for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients' age will be ranged between 30-50 years.
* Both genders will participate in this study.
* All patients suffering from shoulder pain and disability following unilateral modified radical NDS or selective NDS.
* All patients will begin the treatment program from 1 to 3 months after NDS.
* All patients will have limited ROM of shoulder flexion, abduction, external rotation.
* All patients enrolled to the study will have their informed consent.

Exclusion Criteria:

* Subjects with rotator cuff tears or other •shoulder ligament injuries.
* Adhesive capsulitis secondary to Diabetes mellitus or fractures.
* Recurrent shoulder dislocation.
* Recent fracture or surgery to the shoulder.
* Reflex sympathetic dystrophy.
* Neurological disorder.
* Epilepsy or any psychological disorders.
* The presence of residual local-regional cancer or distant metastases to other regions.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Digital Goniometer | 2 months
  Digital goniometer is a device which measures joint ranges, together with velocity and acceleration variables, with a high level of precision and at a relatively low-cost, practically similar to current analogical tools. The digital goniometer is a device specifically designed for the measurement of angles of movement of the human body with a resolution of 1°, representing an ideal substitute to traditional goniometers, which are usually based on a scale of 5° increments

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index | 2 months
  The shoulder pain and disability index (SPADI) is a self-report questionnaire developed to measure the pain and disability associated with shoulder pathology. The SPADI consists of 13 items in two subscales: pain (5 items) and disability (8 items), the original version has each item scored on a visual analogue scale (VAS) and a second version has items scored on a numerical rating scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethical Committee Faculty of Physical Therapy, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt